CLINICAL TRIAL: NCT06675656
Title: Predictive Role of Microbiome in Patients With Urothelial Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo Alfano, PhD, IRCCS San Raffaele
Other Study IDs: UROBIOTA
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1M. Predictive role of microbiome in male with low grade NMIBC undergoing Gem/Dox.: Predictive role of microbiome in male with low grade non-muscle invasive bladder carcinoma undergoing Gem/Dox.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.
- 1F. Predictive role of microbiome in female with low grade NMIBC undergoing Gem/Dox.: Predictive role of microbiome in female with low grade non-muscle invasive bladder carcinoma undergoing Gem/Dox.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.
- 2M. Predictive role of microbiome in male with intermediate grade NMIBC undergoing MMC.: Predictive role of microbiome in male with intermediate grade non-muscle invasive bladder carcinoma undergoing MMC.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.
- 2F. Predictive role of microbiome in female with intermediate grade NMIBC undergoing MMC.: Predictive role of microbiome in female with intermediate grade non-muscle invasive bladder carcinoma undergoing MMC.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.
- 3M. Predictive role of microbiome in male with high grade NMIBC undergoing BCG.: Predictive role of microbiome in male with high grade non-muscle invasive bladder carcinoma undergoing BCG.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.
- 3F. Predictive role of microbiome in female with high grade NMIBC undergoing BCG.: Predictive role of microbiome in female with high grade non-muscle invasive bladder carcinoma undergoing BCG.
  Interventions: Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood.

INTERVENTIONS:
Other: DNA extraction from urine, stool and biopsy. Isolation of serum and PBMC from peripheral blood. — DNA extraction from urine, stool and biopsy for microbiome analysis. Isolation of peripheral blood mononuclear cells from peripheral blood for immunophenotypic analysis, and isolation of serum for analysis of cytokines and bacterial metabolites.

SUMMARY:
This study aims to establish the microbiota composition as a predictive tool for the response to the intravesical immunotherapy with Bacillus Calmette-Guérin (BCG) and 2 different chemotherapies schemes.

In this prospective cohort study patients with low/intermediate/high risk non muscle invasive bladder carcinoma (NMIBC) that undergo BCG/chemo treatment will be enrolled to collect urine stool and blood at different endpoints. Microbiota, short-chain fatty acids and immunophenotype will be quantified to develop a predictive screening platform, which might also integrate traditional urinary cytology and FISH data.

DETAILED DESCRIPTION:
The purpose of this research is to understand the possible use of microbial profile from catheterized urine and feces of patients with NMIBC to categorize patients in two groups: those likely to respond positively and those unlikely to respond to the therapy. Goal of this study is to identify the predictive role of the microbiome to therapy response, thus allowing clinicians to deliver the most appropriate treatment based on the microbiome (microbiome-personalized therapy).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years, all able to signed informed consent form;
* Diagnosis of NMIBC provided by an experience pathology, by using tissue specimens that were staged according to the TNM classification and morphoarchitectural criteria according to the WHO classification.

Exclusion Criteria:

* Participants with ongoing urinary tract infection;
* Antibiotic treatment within the last month;
* Immuno-/chemo- therapy within the past 3 months;
* Chronic immunosuppressive therapy;
* Additional major diagnosis known to affect the gut or bladder microbiota;
* Use of probiotics;
* Uncontrolled diabetes;
* Participants with other malignancy or previous history of oncological or autoimmune diseases.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosis of NMIBC, both first diagnosis or relapsing NMIBC.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Establish the change of microbial profile in high-grade NMIBC patients after BCG administration | 2 years
  Establish the change of urinary and fecal microbiome richness and diversity, and immunophenotype in bladder carcinoma patients after intravesical BCG treatment.

SECONDARY OUTCOMES:
The predictive role of microbiome in BCG responsiveness | 11 years
  Categorize potential candidates for BCG therapy, based on the microbiota pre-therapy.